CLINICAL TRIAL: NCT02887677
Title: A Study of the Effects of Dapagliflozin on Ambulatory Aortic Pressure, Arterial Stiffness and Urine Albumin Excretion in Patients With Type 2 Diabetes
Brief Title: Effects of Dapagliflozin on Central Hemodynamics and Urine Albumin Excretion in Patients With Type 2 Diabetes.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: On February 2019 Astra-Zeneca Greece decided to stop the financial support of the study.
Sponsor: Hellenic Society for Medical Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ESR-15-10964
Record Dates: First submitted 2016-08-25; First posted 2016-09-02 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus
Keywords: Dapagliflozin; Arterial Stiffness; Aortic Pressure
MeSH Terms: conditions — Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dapagliflozin (Active Comparator): Dapagliflozin for oral administration. Patients will be randomized in a 1:1 ratio to the dapagliflozin or placebo group.
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Placebo for oral administration. Patients will be randomized in a 1:1 ratio to the dapagliflozin or placebo group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Administration of dapagliflozin (film-coated tablet of 10mg, per os, q24h, 12 weeks)
  Other Names: Forxiga
  Arms: Dapagliflozin
Drug: Placebo — Administration of placebo (film-coated tablet of same color and texture with dapagliflozin, 10mg, per os, q24h, 12 weeks).
  Arms: Placebo

SUMMARY:
This study is designed to test the hypothesis that the treatment-induced reductions in the ambulatory aortic pressure are more pronounced in the group of dapagliflozin than in the group of placebo.

It is a 12 week, double-blind, randomized, placebo-controlled clinical trial of dapagliflozin versus placebo in 160 adult patients with type 2 diabetes mellitus (DM). It will be conducted in three centers.

Potentially eligible patients will be asked to provide written informed consent (Screening Visit). Patients, who fulfill the inclusion and exclusion criteria, will be asked to visit the sites one week (Visit 1 - V1) after the screening visit. On Visit 2 (V2) all eligible patients will be randomized to one of the two treatment arms and will continue with the next visits as appropriate (Visit 3, Telephone Visit 1, Visit 4-end of study).

Aortic blood pressure (BP) and arterial stiffness parameters will be measured as indicated by the protocol in V1 and V3 with the Mobil-O-Graph monitor.

Blood samples will be collected as indicated by the protocol in Screening Visit for the measurement of glycated hemoglobin (HbA1c), creatinine and liver function parameters. In addition, blood samples will be collected in V1 and V3 for routine hematological and biochemical tests including creatinine, fasting glucose, HbA1c, lipid profile and liver function parameters.

Urine samples will be collected as indicated by the protocol in V1 and V3 for the measurement of albumin to creatinine ratio.

DETAILED DESCRIPTION:
Study design

Screening visit: Potentially eligible patients will be asked to provide written informed consent. The investigators will record full medical history, clinical examination, demographic characteristics, electrocardiogram (ECG), body weight, height, body mass index (BMI) and waist perimeter. Office blood pressure (BP) will be measured by the physicians three times using a mercury sphygmomanometer [cuffs will be placed at the level of brachial artery and a three minute interval will intercept each measurement, following 10 minutes of rest in the seated position (the cuff will cover at least 80% of the brachial circumference and 2/3 of the brachial length.)]. The investigators will also collect blood samples to determine glycated hemoglobin (HbA1C), creatinine, glomerular filtration rate (GFR) and liver function.

Visit 1 (V1): Patients, who fulfill the inclusion and exclusion criteria, will be asked to visit the sites 1 week after the screening visit (+/-2 days), following a 12-hour fast. Three measurements of office BP at the level of brachial artery, with a three minutes interval between each measurement, will be performed with the use of a mercury sphygmomanometer, after 10 minutes-rest in the sitting posture (cuff with bladder size encircling at least 80% of arm circumference and covering two thirds of arm length). After that, venous blood specimens and a spot urine specimen will be collected for relevant blood tests and albumin/creatinine ratio (ACR) respectively. Subsequently, the Mobil-O-Graph monitor with a cuff of appropriate size will be fitted and the BP recording will be initiated for 24 hours. The device will be programmed to collect data every 20 minutes, except for 23:00 to 07:00 (data collection every 30 minutes).

Visit 2 (V2): An appointment will be scheduled the following day for the patient to drop-off the Mobil-O-Graph device. Patients will be randomized in a 1:1 ratio to the dapagliflozin or placebo group and will start receiving the drug regimen the same day. Moreover, all patients will receive dietary and lifestyle advice commencing from this visit.

Telephone Visit 1 (ΤV1): A telephone visit (TV1) will be scheduled 6 weeks after V2 (+/-2 days). Patient history will be obtained, emphasizing on possible adverse events during the previous 6 weeks. Home blood glucose levels, if available, would be also discussed.

Visit 3 (V3): Visit 3 will be scheduled 6 weeks after telephone visit 1 (TV1) (+/-2 days). The following parameters will be determined: medical history of the last weeks, clinical examination (including three brachial BP measurements with a mercury sphygmomanometer as mentioned before), venous blood specimen collection (under 12-hour fast) and the initiation of 24-hour ambulatory blood pressure monitoring (ABPM) (Mobil-O-Graph device). The patients will also provide a spot urine specimen for ACR evaluation.

Visit 4 (V4): Visit 4 will be scheduled 1 day after visit 3. Patients will drop-off the Mobil-O-Graph device.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 and ≤75 years old
* Type 2 diabetes mellitus
* Glycated hemoglobin ≥7% and ≤ 9%
* Patients on monotherapy or combination of two of the following type of antidiabetic agents :metformin, sulphonylurea,DPP-4 inhibitor,or insulin for the past 3 months.
* Patient to provide informed consent

Exclusion Criteria:

* Hypovolemic patients.
* Patients on loop diuretics.
* Patients with low BP (office SBP <110 mmHg) or orthostatic hypotension (BP drop >20 mmHg and SBP <110 mmHg in standing position at 1 min).
* Patients on GLP-1 receptor agonist or pioglitazone.
* Secondary hypertension.
* Stage 2 hypertension or higher (office SBP ≥160 mmHg or DBP ≥100 mmHg).
* Chronic kidney disease stage 3 or higher (GFR<60 mL/min/1.73 m2).
* Myocardial infarction or unstable angina episode within the past 3 months, or congestive heart failure class III-IV according to New York Heart Association criteria.
* Pregnancy or childbearing potential [defined as women which have entered menses and are not post-menopausal (menopause is defined as the absence of menses for at least 12 months without any other medical cause in women of typical age) or women that have been subjected to permanent sterilization (ie. tubal ligation, hysterectomy, bilateral oophorectomy or bilateral salpingectomy)].
* History of liver disease or significant abnormal liver function defined as aspartate aminotransferase (AST) >3x upper limit of normal (ULN) and/or alanine aminotransferase (ALT) >3x ULN or total bilirubin >2.0 mg/dL.
* History of malignancy of any organ system (resected basal cell carcinoma considered cured is exempted) within the past 5 years prior to Visit 1 (V1).
* History of drug or alcohol abuse within the last one year.
* Any contraindication or history of hypersensitivity to the study drug or to drugs with similar chemical structures.
* Any other surgical or medical condition that, in the opinion of the investigator, place the patient at higher risk from his/her participation in the study, or are likely to prevent the patient from complying with the requirements of the study or completing the trial period.
* Intake of an investigational drug in another trial within 30 days prior to Visit 1 (V1).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Ambulatory systolic aortic pressure | 12 weeks

SECONDARY OUTCOMES:
Ambulatory aortic (central) diastolic blood pressure (DBP) | 12 weeks
Ambulatory brachial systolic blood pressure (SBP) and DBP | 12 weeks
Ambulatory augmentation index (AIx) | 12 weeks
Ambulatory pulse wave velocity (PWV) | 12 weeks
Office brachial SBP and DBP | 12 weeks
Albumin/creatinine ratio (ACR) | 12 weeks
Lipid profile (Total-Cholesterol, LDL-Cholesterol, HDL-Cholesterol, triglycerides) | 12 weeks
HbA1c | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pantelis Sarafidis, Principal Investigator — Aristotle University Of Thessaloniki
Locations (3):
- Greece (3):
  - Ahepa Hospital, Thessaloniki
  - Hippokrateio Hospital, Thessaloniki
  - Papageorgiou Hospital, Thessaloniki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shaw JE, Sicree RA, Zimmet PZ. Global estimates of the prevalence of diabetes for 2010 and 2030. Diabetes Res Clin Pract. 2010 Jan;87(1):4-14. doi: 10.1016/j.diabres.2009.10.007. Epub 2009 Nov 6. PMID 19896746
- [Background] Hu FB. Globalization of diabetes: the role of diet, lifestyle, and genes. Diabetes Care. 2011 Jun;34(6):1249-57. doi: 10.2337/dc11-0442. PMID 21617109
- [Background] Martin-Timon I, Sevillano-Collantes C, Segura-Galindo A, Del Canizo-Gomez FJ. Type 2 diabetes and cardiovascular disease: Have all risk factors the same strength? World J Diabetes. 2014 Aug 15;5(4):444-70. doi: 10.4239/wjd.v5.i4.444. PMID 25126392
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Abdul-Ghani MA, Norton L, DeFronzo RA. Efficacy and safety of SGLT2 inhibitors in the treatment of type 2 diabetes mellitus. Curr Diab Rep. 2012 Jun;12(3):230-8. doi: 10.1007/s11892-012-0275-6. PMID 22528597
- [Background] Aylsworth A, Dean Z, VanNorman C, Nkemdirim Okere A. Dapagliflozin for the Treatment of Type 2 Diabetes Mellitus. Ann Pharmacother. 2014 Sep;48(9):1202-1208. doi: 10.1177/1060028014540450. Epub 2014 Jun 20. PMID 24951310
- [Background] Defronzo RA. Banting Lecture. From the triumvirate to the ominous octet: a new paradigm for the treatment of type 2 diabetes mellitus. Diabetes. 2009 Apr;58(4):773-95. doi: 10.2337/db09-9028. No abstract available. PMID 19336687
- [Background] Karagiannis A, Tziomalos K, Anagnostis P, Gossios TD, Florentin M, Athyros VG, Mikhailidis DP. The effect of antihypertensive agents on insulin sensitivity, lipids and haemostasis. Curr Vasc Pharmacol. 2010 Nov;8(6):792-803. doi: 10.2174/157016110793563906. PMID 20626344
- [Background] Inzucchi SE, Bergenstal RM, Buse JB, Diamant M, Ferrannini E, Nauck M, Peters AL, Tsapas A, Wender R, Matthews DR; American Diabetes Association (ADA); European Association for the Study of Diabetes (EASD). Management of hyperglycemia in type 2 diabetes: a patient-centered approach: position statement of the American Diabetes Association (ADA) and the European Association for the Study of Diabetes (EASD). Diabetes Care. 2012 Jun;35(6):1364-79. doi: 10.2337/dc12-0413. Epub 2012 Apr 19. No abstract available. PMID 22517736
- [Background] Pandey R, Kumar N, Yadav M, Nagpal R, Jain S, Yadav H. Anti-diabetic compounds and their patent information: an update. Recent Pat Inflamm Allergy Drug Discov. 2013 Jan 1;7(1):35-48. PMID 23016523
- [Background] Karagiannis T, Paschos P, Paletas K, Matthews DR, Tsapas A. Dipeptidyl peptidase-4 inhibitors for treatment of type 2 diabetes mellitus in the clinical setting: systematic review and meta-analysis. BMJ. 2012 Mar 12;344:e1369. doi: 10.1136/bmj.e1369. PMID 22411919
- [Background] Hoerger TJ, Segel JE, Gregg EW, Saaddine JB. Is glycemic control improving in U.S. adults? Diabetes Care. 2008 Jan;31(1):81-6. doi: 10.2337/dc07-1572. Epub 2007 Oct 12. PMID 17934153
- [Background] Xu X, Wang G, Zhou T, Chen L, Chen J, Shen X. Novel approaches to drug discovery for the treatment of type 2 diabetes. Expert Opin Drug Discov. 2014 Sep;9(9):1047-58. doi: 10.1517/17460441.2014.941352. Epub 2014 Jul 23. PMID 25054271
- [Background] Tasyurek HM, Altunbas HA, Balci MK, Sanlioglu S. Incretins: their physiology and application in the treatment of diabetes mellitus. Diabetes Metab Res Rev. 2014 Jul;30(5):354-71. doi: 10.1002/dmrr.2501. PMID 24989141
- [Background] DeFronzo RA, Davidson JA, Del Prato S. The role of the kidneys in glucose homeostasis: a new path towards normalizing glycaemia. Diabetes Obes Metab. 2012 Jan;14(1):5-14. doi: 10.1111/j.1463-1326.2011.01511.x. PMID 21955459
- [Background] Wright EM, Turk E. The sodium/glucose cotransport family SLC5. Pflugers Arch. 2004 Feb;447(5):510-8. doi: 10.1007/s00424-003-1063-6. Epub 2003 May 14. PMID 12748858
- [Background] Vlotides G, Mertens PR. Sodium-glucose cotransport inhibitors: mechanisms, metabolic effects and implications for the treatment of diabetic patients with chronic kidney disease. Nephrol Dial Transplant. 2015 Aug;30(8):1272-6. doi: 10.1093/ndt/gfu299. Epub 2014 Sep 17. PMID 25230708
- [Background] Chao EC, Henry RR. SGLT2 inhibition--a novel strategy for diabetes treatment. Nat Rev Drug Discov. 2010 Jul;9(7):551-9. doi: 10.1038/nrd3180. Epub 2010 May 28. PMID 20508640
- [Background] Rahmoune H, Thompson PW, Ward JM, Smith CD, Hong G, Brown J. Glucose transporters in human renal proximal tubular cells isolated from the urine of patients with non-insulin-dependent diabetes. Diabetes. 2005 Dec;54(12):3427-34. doi: 10.2337/diabetes.54.12.3427. PMID 16306358
- [Background] Rosenwasser RF, Sultan S, Sutton D, Choksi R, Epstein BJ. SGLT-2 inhibitors and their potential in the treatment of diabetes. Diabetes Metab Syndr Obes. 2013 Nov 27;6:453-67. doi: 10.2147/DMSO.S34416. PMID 24348059
- [Background] Albarran OG, Ampudia-Blasco FJ. [Dapagliflozin, the first SGLT-2 inhibitor in the treatment of type 2 diabetes]. Med Clin (Barc). 2013 Sep;141 Suppl 2:36-43. doi: 10.1016/S0025-7753(13)70062-9. Spanish. PMID 24444523
- [Background] Sun YN, Zhou Y, Chen X, Che WS, Leung SW. The efficacy of dapagliflozin combined with hypoglycaemic drugs in treating type 2 diabetes mellitus: meta-analysis of randomised controlled trials. BMJ Open. 2014 Apr 7;4(4):e004619. doi: 10.1136/bmjopen-2013-004619. PMID 24710132
- [Background] Vasilakou D, Karagiannis T, Athanasiadou E, Mainou M, Liakos A, Bekiari E, Sarigianni M, Matthews DR, Tsapas A. Sodium-glucose cotransporter 2 inhibitors for type 2 diabetes: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 20;159(4):262-74. doi: 10.7326/0003-4819-159-4-201308200-00007. PMID 24026259
- [Background] Sarafidis PA, Georgianos PI, Lasaridis AN. Diuretics in clinical practice. Part I: mechanisms of action, pharmacological effects and clinical indications of diuretic compounds. Expert Opin Drug Saf. 2010 Mar;9(2):243-57. doi: 10.1517/14740330903499240. PMID 20095917
- [Background] Sarafidis PA, Bakris GL. State of hypertension management in the United States: confluence of risk factors and the prevalence of resistant hypertension. J Clin Hypertens (Greenwich). 2008 Feb;10(2):130-9. doi: 10.1111/j.1751-7176.2008.07309.x. PMID 18256578
- [Background] Bakris G, Molitch M, Hewkin A, Kipnes M, Sarafidis P, Fakouhi K, Bacher P, Sowers J; STAR Investigators. Differences in glucose tolerance between fixed-dose antihypertensive drug combinations in people with metabolic syndrome. Diabetes Care. 2006 Dec;29(12):2592-7. doi: 10.2337/dc06-1373. PMID 17130190
- [Background] Ferrannini E, Ramos SJ, Salsali A, Tang W, List JF. Dapagliflozin monotherapy in type 2 diabetic patients with inadequate glycemic control by diet and exercise: a randomized, double-blind, placebo-controlled, phase 3 trial. Diabetes Care. 2010 Oct;33(10):2217-24. doi: 10.2337/dc10-0612. Epub 2010 Jun 21. PMID 20566676
- [Background] Wilding JP, Woo V, Soler NG, Pahor A, Sugg J, Rohwedder K, Parikh S; Dapagliflozin 006 Study Group. Long-term efficacy of dapagliflozin in patients with type 2 diabetes mellitus receiving high doses of insulin: a randomized trial. Ann Intern Med. 2012 Mar 20;156(6):405-15. doi: 10.7326/0003-4819-156-6-201203200-00003. PMID 22431673
- [Background] Nauck MA, Del Prato S, Duran-Garcia S, Rohwedder K, Langkilde AM, Sugg J, Parikh SJ. Durability of glycaemic efficacy over 2 years with dapagliflozin versus glipizide as add-on therapies in patients whose type 2 diabetes mellitus is inadequately controlled with metformin. Diabetes Obes Metab. 2014 Nov;16(11):1111-20. doi: 10.1111/dom.12327. Epub 2014 Jul 10. PMID 24919526
- [Background] Karagiannis A, Hatzitolios AI, Athyros VG, Deligianni K, Charalambous C, Papathanakis C, Theodosiou G, Drakidis T, Chatzikaloudi V, Kamilali C, Matsiras S, Matziris A, Savopoulos C, Baltatzi M, Rudolf J, Tziomalos K, Mikhailidis DP. Implementation of guidelines for the management of arterial hypertension. The impulsion study. Open Cardiovasc Med J. 2009 May 5;3:26-34. doi: 10.2174/1874192400903010026. PMID 19557149
- [Background] Gorostidi M, Vinyoles E, Banegas JR, de la Sierra A. Prevalence of white-coat and masked hypertension in national and international registries. Hypertens Res. 2015 Jan;38(1):1-7. doi: 10.1038/hr.2014.149. Epub 2014 Oct 16. PMID 25319601
- [Background] Clement DL, De Buyzere ML, De Bacquer DA, de Leeuw PW, Duprez DA, Fagard RH, Gheeraert PJ, Missault LH, Braun JJ, Six RO, Van Der Niepen P, O'Brien E; Office versus Ambulatory Pressure Study Investigators. Prognostic value of ambulatory blood-pressure recordings in patients with treated hypertension. N Engl J Med. 2003 Jun 12;348(24):2407-15. doi: 10.1056/NEJMoa022273. PMID 12802026
- [Background] Weber MA, Mansfield TA, Alessi F, Iqbal N, Parikh S, Ptaszynska A. Effects of dapagliflozin on blood pressure in hypertensive diabetic patients on renin-angiotensin system blockade. Blood Press. 2016;25(2):93-103. doi: 10.3109/08037051.2015.1116258. Epub 2015 Dec 1. PMID 26623980
- [Background] Weber MA, Mansfield TA, T'joen C, Ptaszynska A (2013) Dapagliflozin for Reduction of Blood Pressure in Diabetic Patients Inadequately Controlled With Combination Antihypertensive Regimen. Circulation, 128; A13165.
- [Background] Lambers Heerspink HJ, de Zeeuw D, Wie L, Leslie B, List J. Dapagliflozin a glucose-regulating drug with diuretic properties in subjects with type 2 diabetes. Diabetes Obes Metab. 2013 Sep;15(9):853-62. doi: 10.1111/dom.12127. Epub 2013 Jun 5. PMID 23668478
- [Background] Vlachopoulos C, Aznaouridis K, O'Rourke MF, Safar ME, Baou K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with central haemodynamics: a systematic review and meta-analysis. Eur Heart J. 2010 Aug;31(15):1865-71. doi: 10.1093/eurheartj/ehq024. Epub 2010 Mar 2. PMID 20197424
- [Background] Tziomalos K, Athyros VG, Karagiannis A. Treating Arterial Stiffness in Young and Elderly Patients with the Metabolic Syndrome. Curr Pharm Des. 2014;20(39):6106-13. doi: 10.2174/1381612820666140417101523. PMID 24745924
- [Background] Jankowski P, Kawecka-Jaszcz K, Czarnecka D, Brzozowska-Kiszka M, Styczkiewicz K, Loster M, Kloch-Badelek M, Wilinski J, Curylo AM, Dudek D; Aortic Blood Pressure and Survival Study Group. Pulsatile but not steady component of blood pressure predicts cardiovascular events in coronary patients. Hypertension. 2008 Apr;51(4):848-55. doi: 10.1161/HYPERTENSIONAHA.107.101725. Epub 2008 Feb 11. PMID 18268136
- [Background] Katsiki N, Koumaras C, Athyros VG, Karagiannis A. Thinking beyond traditional cardiovascular risk factors: the role of arterial stiffness in targeting residual risk. Angiology. 2012 Jan;63(1):9-11. doi: 10.1177/0003319711406256. No abstract available. PMID 22144689
- [Background] Koumaras C, Tzimou M, Stavrinou E, Griva T, Gossios TD, Katsiki N, Athyros VG, Mikhailidis DP, Karagiannis A. Role of antihypertensive drugs in arterial 'de-stiffening' and central pulsatile hemodynamics. Am J Cardiovasc Drugs. 2012 Jun 1;12(3):143-56. doi: 10.2165/11599040-000000000-00000. PMID 22540323
- [Background] Vlachopoulos C, Aznaouridis K, Stefanadis C. Prediction of cardiovascular events and all-cause mortality with arterial stiffness: a systematic review and meta-analysis. J Am Coll Cardiol. 2010 Mar 30;55(13):1318-27. doi: 10.1016/j.jacc.2009.10.061. PMID 20338492
- [Background] Wassertheurer S, Kropf J, Weber T, van der Giet M, Baulmann J, Ammer M, Hametner B, Mayer CC, Eber B, Magometschnigg D. A new oscillometric method for pulse wave analysis: comparison with a common tonometric method. J Hum Hypertens. 2010 Aug;24(8):498-504. doi: 10.1038/jhh.2010.27. Epub 2010 Mar 18. PMID 20237499
- [Background] Protogerou AD, Argyris A, Nasothimiou E, Vrachatis D, Papaioannou TG, Tzamouranis D, Blacher J, Safar ME, Sfikakis P, Stergiou GS. Feasibility and reproducibility of noninvasive 24-h ambulatory aortic blood pressure monitoring with a brachial cuff-based oscillometric device. Am J Hypertens. 2012 Aug;25(8):876-82. doi: 10.1038/ajh.2012.63. Epub 2012 Jun 7. PMID 22673021
- [Background] Sarafidis PA, Georgianos PI, Karpetas A, Bikos A, Korelidou L, Tersi M, Divanis D, Tzanis G, Mavromatidis K, Liakopoulos V, Zebekakis PE, Lasaridis A, Protogerou AD. Evaluation of a novel brachial cuff-based oscillometric method for estimating central systolic pressure in hemodialysis patients. Am J Nephrol. 2014;40(3):242-50. doi: 10.1159/000367791. Epub 2014 Oct 11. PMID 25322847
- [Background] Parati G, Stergiou G, O'Brien E, Asmar R, Beilin L, Bilo G, Clement D, de la Sierra A, de Leeuw P, Dolan E, Fagard R, Graves J, Head GA, Imai Y, Kario K, Lurbe E, Mallion JM, Mancia G, Mengden T, Myers M, Ogedegbe G, Ohkubo T, Omboni S, Palatini P, Redon J, Ruilope LM, Shennan A, Staessen JA, vanMontfrans G, Verdecchia P, Waeber B, Wang J, Zanchetti A, Zhang Y; European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. European Society of Hypertension practice guidelines for ambulatory blood pressure monitoring. J Hypertens. 2014 Jul;32(7):1359-66. doi: 10.1097/HJH.0000000000000221. PMID 24886823
- [Background] Weber T, Wassertheurer S, Rammer M, Maurer E, Hametner B, Mayer CC, Kropf J, Eber B. Validation of a brachial cuff-based method for estimating central systolic blood pressure. Hypertension. 2011 Nov;58(5):825-32. doi: 10.1161/HYPERTENSIONAHA.111.176313. Epub 2011 Sep 12. PMID 21911710
- [Background] Papaioannou TG, Argyris A, Protogerou AD, Vrachatis D, Nasothimiou EG, Sfikakis PP, Stergiou GS, Stefanadis CI. Non-invasive 24 hour ambulatory monitoring of aortic wave reflection and arterial stiffness by a novel oscillometric device: the first feasibility and reproducibility study. Int J Cardiol. 2013 Oct 25;169(1):57-61. doi: 10.1016/j.ijcard.2013.08.079. Epub 2013 Sep 8. PMID 24063914
- [Background] Franssen PM, Imholz BP. Evaluation of the Mobil-O-Graph new generation ABPM device using the ESH criteria. Blood Press Monit. 2010 Aug;15(4):229-31. doi: 10.1097/mbp.0b013e328339be38. PMID 20658764
- [Background] Wei W, Tolle M, Zidek W, van der Giet M. Validation of the mobil-O-Graph: 24 h-blood pressure measurement device. Blood Press Monit. 2010 Aug;15(4):225-8. doi: 10.1097/MBP.0b013e328338892f. PMID 20216407
- [Background] Laurent S, Cockcroft J, Van Bortel L, Boutouyrie P, Giannattasio C, Hayoz D, Pannier B, Vlachopoulos C, Wilkinson I, Struijker-Boudier H; European Network for Non-invasive Investigation of Large Arteries. Expert consensus document on arterial stiffness: methodological issues and clinical applications. Eur Heart J. 2006 Nov;27(21):2588-605. doi: 10.1093/eurheartj/ehl254. Epub 2006 Sep 25. PMID 17000623
- [Background] Hametner B, Wassertheurer S, Kropf J, Mayer C, Eber B, Weber T. Oscillometric estimation of aortic pulse wave velocity: comparison with intra-aortic catheter measurements. Blood Press Monit. 2013 Jun;18(3):173-6. doi: 10.1097/MBP.0b013e3283614168. PMID 23571229
- [Background] Protogerou AD, Smulyan H, Safar ME. Closer to noninvasive out-of-office aortic blood pressure assessment: a time to think and act. Hypertension. 2011 Nov;58(5):765-7. doi: 10.1161/HYPERTENSIONAHA.111.177501. Epub 2011 Sep 12. No abstract available. PMID 21911711
- [Derived] Papadopoulou E, Theodorakopoulou MP, Loutradis C, Tzanis G, Tzatzagou G, Kotsa K, Zografou I, Tsapas A, Karagiannis A, Sarafidis P. Dapagliflozin Does Not Affect Short-Term Blood Pressure Variability in Patients With Type 2 Diabetes Mellitus. Am J Hypertens. 2021 Apr 20;34(4):404-413. doi: 10.1093/ajh/hpaa207. PMID 33277990